CLINICAL TRIAL: NCT04056598
Title: Characterization of Immune Responses Against Acne-associated Bacterium Propionibacterium Acnes - a Pilot Study
Brief Title: Acne Vulgaris Related Microbiology and Serology
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Collaborators: CRAT (Unknown)
Responsible Party: Sponsor
Other Study IDs: SAIRB-17-0087
Record Dates: First submitted 2019-08-05; First posted 2019-08-14 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Acne Vulgaris
Keywords: P. acnes; acne vulgaris; humoral immune response; microbiome; SLST
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Patient serum samples and facial swabs for microbiome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate to severe acne vulgaris: Determined by the acne severity grade of IGA 2 and above
  Interventions: Diagnostic Test: Study of humoral immunity
- Mild acne vulgaris: Determined by the severity grade of IGA <2
  Interventions: Diagnostic Test: Study of humoral immunity

INTERVENTIONS:
Diagnostic Test: Study of humoral immunity — Analysis: Surface antigen ELISA, recognition of living P. acnes bacteria via FACS, 16SRNA study of microbiome, SLST typing of P. acnes bacteria
  Other Names: Study of skin microbiome

SUMMARY:
This will be an investigation to determine the quality of the serological immune responses against Propionibacterium acnes (P. acnes) in acne patients compared to healthy individuals. In particular, the investigators will measure serum antibody titers against P. acnes surface antigens, and the efficiency of antibody-mediated phagocytic killing of P. acnes.

DETAILED DESCRIPTION:
Acne vulgaris, which affects >85% of teenagers and >10% of adults, was recently re-defined as a complex chronic disease associated with Propionibacterium acnes (P. acnes). Until recently, the pathogenic role of bacteria Propionibacterium acnes (P. acnes) has been debated due to the fact that this bacterium is also found, although in lower density, on the skin of healthy individuals. However, in the last few years, genomic sequencing and the comparative analysis of >250 P. acnes strains revealed the existence of the strains prevalently associated with severe cases of acne. In the study that analyzed more than 200 clinical isolates, it was found that 75% of the P. acnes strains that were isolated from acne lesions of acne patients, belonged to genetic type I-IA and that this group also represented 85% of the antibiotic resistant P. acnes strains isolated in the course of the study. This provided the first clear evidence for the virulent potential of P. acnes, that has been previously suspected also in some cases of eye, bone and post-operative infections. More recent research studies have identified additional virulent strains which can be distinguished based on the ribosomal DNA analysis.

Although these genetic studies have revealed the existence of virulent P. acnes strains, it is not yet clear how these strains promote disease pathogenesis and symptoms, and whether the host immune response either exaggerates or ameliorates the disease. In particular, there have been no systematic studies regarding the role of a central immunity in the protection against this pathogen.

Therefore, this will be one of the first studies to address scientifically and therapeutically important questions including:

1. Immunogenicity of P. acnes in the acne patients compared to healthy individuals who are recovered from moderate or severe acne vulgaris.
2. The role of antibodies in controlling colonization and acne development due to P. acnes
3. The relationship between P. acnes genetic information and serotype classification, based on the immune recognition pattern (the degree of the similarity among genetically different strains based on the surface components recognition by the immune system) Answering these questions could support development of novel and better treatment options, which could significantly improve the outcome in acne vulgaris patients. Existing acne treatments either treat the symptoms only on skin surface (e.g. topical agents: creams, lotions), or are not offering long-term solutions (antibiotics, vitamin A derivatives). Moreover, antibiotics raise antibiotic resistance among P. acnes as well as other types of bacteria and increase the risk of super-infection by other pathogens. Vitamin A derivatives are not effective in all patients and post-therapy relapse is common; besides, they are not routinely prescribed to patients due to serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Acne patients (18 - 40 years of age)
* Clinical diagnosis of medium acne vulgaris (covering more than 30% of the patient's face and loaded with comedones, pustules and acne lesions of >2 cm in size) for at least six months or longer
* Clinical diagnosis of severe acne vulgaris (acne conglobata, sinus or cystic type acne covering most of the face (>60% of the facial surface) - IGA 3-4) for at least six months or longer
* Age-matched healthy adults (between 18 and 40 years), with history of moderate or severe acne, but who have been free from acne for more than two years - 'free from acne' period may include minor, intermittent breakouts due to hormonal reasons, such as menstruation

Exclusion Criteria:

* Subjects who received anti-acne antibiotic therapy less than 2 months prior to recruitment
* Subjects who received isotretinoin therapy within the last 6 months
* Subjects who were using hormonal contraceptives within the last 3 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects for the study will be drawn from:
  * Study group: Acne patients, 18-40 years of age, currently suffering from moderate or severe acne vulgaris
  * Control group: Healthy individuals of 18-40 years of age, who recovered from moderate or severe acne vulgaris
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation of acne vulgaris severity with humoral immunity assessed by ELISA, binding to P. acnes strains and OPK assay | Serum samples will be collected at visit and samples will be investigated upon availability of all samples. Analysis will occur an average of 1 year and will reflect patient's immune status at visit.
  Quantitative and qualitative investigation of serum immuno globulins by (1) P. acnes surface antigen specific ELISA (EC50), (2) FACS binding (MFI) analysis on living P. acnes microorganisms of the most relevant SLST's and (3) opsono-phagocytotic killing potency (% killing) on the most important P. acnes strains in presence of human effector cells
Correlation of acne vulgaris severity with skin microbiome identified in acne lesions and by facial swabs | Swabs will be collected at visit and samples will be investigated upon availability of all samples. Analysis will be done an average of 1 year and will reflect patient's microbiome (on skin and in acne lesions) at visit.
  Swabs from skin (cheak and front head) and acne lesions (pustules) will be collected and microbiome (presence of specific microorganism) will be analyzed by NGS. SLST (SLST typing) will be applied to characterize in detail identified P. acnes strains

SECONDARY OUTCOMES:
Correlation of microbiome identified on skin and acne lesion samples (Outcome 2) with humoral immunity (Outcome 1) | Serum and microbiome samples will be collected at patient's visit. Analysis will be done an average of 1 year and will reflect patient status at visit.
  We will investigate a potential correlation between results from assessment of humoral immunity (Outcome 1) and patient specific microbiome identified in skin lesions and on the skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Associates of Tidewater, Norfolk, Virginia, United States